CLINICAL TRIAL: NCT05523453
Title: Examination and Refinement of a Novel Treatment for Posttraumatic Stress Disorder: Processing of Positive Memories Technique (PPMT)
Brief Title: Examining Effects of a Therapeutic Focus on Positive Memories on Post-Trauma Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Responsible Party: Principal Investigator, Ateka Contractor, Associate Professor, University of North Texas, Denton, TX
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R15MH129773-01A1 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-08-31 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stress Disorders, Post-Traumatic; Affect; Memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Processing of Positive Memories Technique (PPMT) (Active Comparator): Participants receive 5 60-minute Processing of Positive Memories Technique (PPMT) sessions for PTSD following the treatment procedures as outlined in PPMT therapy manual.
  Interventions: Behavioral: Processing of Positive Memories Technique (PPMT)
- Supportive Counseling (SC) (Active Comparator): Participants receive 5 60-minute supportive counseling (SC) sessions. SC includes a discussion of the daily monitoring diary and exploration of current issues and concerns.
  Interventions: Behavioral: Supportive Counseling (SC)

INTERVENTIONS:
Behavioral: Processing of Positive Memories Technique (PPMT) — PPMT comprises of 5 sessions focused on identifying and processing positive memories. In Session 1-5, participants narrate details of one positive memory, and process the positive memory to elicit positive values, affect, strengths, and thoughts.
  Arms: Processing of Positive Memories Technique (PPMT)
Behavioral: Supportive Counseling (SC) — SC is a 5-session, active and non-specific treatment administered weekly, which includes a discussion of the daily monitoring diary and exploration of current issues and concerns.
  Arms: Supportive Counseling (SC)

SUMMARY:
Posttraumatic stress disorder (PTSD) has devastating health consequences. Evidence-based PTSD interventions address the substantial burden of PTSD on the health of individuals and societies; however, several individuals receiving these interventions drop out and not all individuals experience improvement in PTSD symptoms. Moreover, these current PTSD interventions primarily target trauma memories. Notably, growing evidence suggests that PTSD symptoms are related to difficulties in the encoding and retrieving of positive memories as well.

Thus, the proposed study will examine effects of and targets underlying a novel PTSD technique focused on narrating and detailing positive memories - Processing of Positive Memories Technique (PPMT). Methodologically, 70 individuals will be randomly assigned to PPMT vs. Supportive Counseling (SC) for this study.

The aims of the proposed study include (1) examining PPMT's effects on PTSD symptom severity and stress systems' dysregulation (i.e., awakening salivary alpha amylase [sAA] and cortisol); (2) examining mechanisms underlying PPMT's effects; and (3) refining PPMT. It is hypothesized that the PPMT arm will report greater decreases in PTSD severity and sAA/cortisol ratios. Further, it is hypothesized that PPMT-related improved affect will mediate the association between study arm (PPMT vs. SC) and changes in PTSD severity. Lastly, feedback will be obtained from study participants on PPMT's feasibility, format, and content to refine PPMT.

The proposed study may contribute preliminary evidence on the potential significance of targeting positive memories in PTSD interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Willing/able to provide informed consent
* Past month DSM-5 posttraumatic stress disorder (PTSD) diagnosis
* Working knowledge of English

Exclusion Criteria:

* Active suicidal intent or attempts
* Active psychosis
* Currently receiving mental health therapy (past 3 months)
* Dosage changes in psychiatric medications (past 3 months)
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Baseline
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Week 1 post-baseline during therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Week 2 post-baseline during therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Week 3 post-baseline during therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Week 4 post-baseline during therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | Week 5 post-baseline during therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | 1 week after last therapy session
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.
Posttraumatic Stress Disorder Checklist for DSM-5 scores | 3-month post treatment completion
  PTSD symptom severity is assessed using 20 items with response options ranging from 0 = not at all to 4 = extremely.

SECONDARY OUTCOMES:
Saliva Samples | 3 times each day for 2 consecutive days prior to first therapy session
  Salivary alpha amylase and cortisol output will be assessed.
Saliva Samples | 3 times each day for 2 consecutive days after the last therapy session
  Salivary alpha amylase and cortisol output will be assessed.
Positive and Negative Affect Schedule | Baseline
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | Week 1 post-baseline during therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | Week 2 post-baseline during therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | Week 3 post-baseline during therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | Week 4 post-baseline during therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | Week 5 post-baseline during therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.
Positive and Negative Affect Schedule | 1 week after last therapy session
  Positive and negative affect is assessed using 20 items with response options ranging from 1 = not at all/very slightly to 5 = extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Ateka Contractor, PHD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Contractor AA, Blumenthal H, Rosenfield D, Shea MT, Taylor DJ, Fentem A, Vingren JL. Study protocol and rationale for a pilot randomized clinical trial comparing processing of positive memories technique with supportive counseling for PTSD. Contemp Clin Trials. 2024 Mar;138:107455. doi: 10.1016/j.cct.2024.107455. Epub 2024 Jan 20. PMID 38253251